CLINICAL TRIAL: NCT00261495
Title: Randomized, Open-Label, Comparative Parallel Group Study to Assess Efficacy and Safety on Flexible Dosages of OROS Hydromorphone Once-Daily Compared to Sustained Release Oxycodone Twice Daily in Subjects With Chronic Non-malignant Pain Requiring Continuous Opioid Therapy.
Brief Title: A Study of the Effectiveness and Safety of Sustained-release Hydromorphone (a Strong Opioid) in Patients With Chronic Noncancer Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002374; OROS-ANA-3001 (Other: Janssen Pharmaceutica N.V.); 2004-005187-24 (EudraCT Number)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: chronic noncancer pain; pain; analgesia; analgesic opioid; oxycodone; hydromorphone
MeSH Terms: conditions — Pain; Agnosia | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone (Active Comparator)
  Interventions: Drug: Oxycodone
- OROS hydromorphone HCl (Experimental)
  Interventions: Drug: OROS hydromorphone HCl

INTERVENTIONS:
Drug: OROS hydromorphone HCl — 8 to 32 mg once daily for 52 weeks (flexible dosing)
  Arms: OROS hydromorphone HCl
Drug: Oxycodone — 10, 20, or 40 mg twice a day for 52 weeks (flexible dosing)
  Arms: Oxycodone

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of sustained- release hydromorphone, formulated to release slowly over time, taken once daily, and controlled- release oxycodone taken twice daily, in patients with chronic non-cancer pain. The study will also determine the dose of sustained-release hydromorphone that provides a level of pain control that is equal to the pain control provided by control-released oxycodone (equi-analgesic dosage).

DETAILED DESCRIPTION:
Conventional immediate-release forms of hydromorphone and oxycodone have a relatively short duration of action that require dosing every 4 to 6 hours. To counterbalance the drawback of repeated opioid intake, sustained-release formulations of oxycodone and hydromorphone were developed that allow twice-daily dosing. Subsequently, a novel, once-daily, extended-release hydromorphone formulation was developed to further enhance ease of treatment and improve effectiveness in the treatment of severe pain. This is a randomized, open-label, comparative, parallel-group, 24-week flexible-dose study in patients with chronic noncancer pain severe enough to require continuous opioid therapy. Patients will receive either 8 mg of sustained-release hydromorphone, taken once daily or 10 mg of controlled-release oxycodone, taken twice daily. Individual adjustments in dosing will be performed to achieve satisfactory pain control, up to a maximum daily dosage of 32 mg for hydromorphone and 80 mg for oxycodone. The primary efficacy outcome will be the determination of the dose of hydromorphone that produces a level of pain control that is equal to the pain control provided by oxycodone (equi-analgesic dose). Safety will be monitored throughout the study. The study hypothesis is that sustained-release hydromorphone taken once daily is well tolerated and is not inferior with regard to pain control to controlled-release oxycodone taken twice daily.

Amendment:

Amendment was made to the duration of the study from duration of '24 weeks' to '52 weeks' in order to collect long-term safety and efficacy data. OROS hydromorphone 8, 16, or 32 mg tablets QD or SR oxycodone 10, 20, or 40 mg tablets BID. Individual adjustments in dosing performed to achieve satisfactory pain control over 24 weeks. Amendment: treatment duration was extended to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic noncancer pain severe enough to require continuous opioid therapy (a score of at least 5 in "pain right now" on a 11 point numeric rating scale) who have never received an opioid or are currently treated with a weak opioid, and who experience insufficient pain control.

Exclusion Criteria:

* Patients who have been treated with strong opioids (including hydromorphone and oxycodone) within the last 4 weeks prior to study inclusion or who will probably undergo any treatment (e.g. neurological techniques, surgery) within the next 6 months, which may abruptly alter degree or nature of pain experienced
* patients with a history of disease(s), current illness, or therapy which would preclude them from participation in the study
* and patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (52):
- Czechia (3):
  - Brno
  - Pilsen
  - Prague
- Denmark (5):
  - Copenhagen
  - Esbjerg
  - Nyborg
  - Svendborg
  - Vejle
- France (4):
  - Amiens
  - Bois-Guillaume
  - Lille
  - Paris
- Germany (18):
  - Berlin
  - Drensteinfurt
  - Dresden
  - Duderstadt
  - Frankfurt
  - Giessen
  - Göppingen
  - Hamburg
  - Herne
  - Jena
  - Kiel
  - Kÿln
  - Ludwigshafen
  - Mannheim
  - Nuremberg
  - Regensburg
  - Rodgau
  - Wiesbaden
- Norway (3):
  - Bodø
  - Lørenskog
  - Oslo
- Poland (5):
  - Gdansk
  - Krakow
  - Lublin
  - Warsaw
  - Wroclaw
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Martin
  - Prešov
- Slovenia (3):
  - Ljubljana
  - Maribor
  - Slovenj Gradec
- Sweden (4):
  - Gothenburg
  - Jönköping
  - Kristianstad
  - Linköping
- Switzerland (3):
  - Aarau
  - Basel
  - Lausanne

REFERENCES:
- [Result] Binsfeld H, Szczepanski L, Waechter S, Richarz U, Sabatowski R. A randomized study to demonstrate noninferiority of once-daily OROS((R)) hydromorphone with twice-daily sustained-release oxycodone for moderate to severe chronic noncancer pain. Pain Pract. 2010 Sep-Oct;10(5):404-15. doi: 10.1111/j.1533-2500.2009.00342.x. PMID 20384968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in 11 countries (Czech Republic, Denmark, France, Germany, Italy, Norway, Poland, Slovakia, Slovenia, Sweden, and Switzerland). 63 study centres randomized subjects and 1 centre screened 1 subject but did not randomize. Recruitment period: 15 March 2006 (first patient in) to 31 March 2007 (last patient in).
Groups:
- OROS Hydromorphone HCl: Initial dose 8 mg (minimum dose), 16 mg, or 32 mg (maximum dose), oral administration, once-daily, 4 weeks (titration phase), 20 weeks (maintenance phase), 28 weeks (extension phase)
- Oxycodone: Initial dose 10 mg (minimum dose), 20 mg, and 40 mg, oral administration, twice daily, 4 weeks (titration phase), 20 weeks (maintenance phase), and 28 weeks (extension phase)
Period: Titration Phase (Weeks 0 to 4)
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Started | 254 | 250
Completed | 206 | 185
Not Completed | 48 | 65
Not completed — Adverse Event | 28 | 36
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Lack of Efficacy | 8 | 8
Not completed — Physician Decision | 3 | 1
Not completed — Non-compliance | 2 | 5
Not completed — Protocol Violation | 1 | 4
Period: Maintenance Phase (Weeks 4 to 24)
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Started | 206 | 185
Completed | 140 | 137
Not Completed | 66 | 48
Not completed — Adverse Event | 29 | 20
Not completed — Lack of Efficacy | 14 | 10
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Non-compliance | 1 | 5
Not completed — Protocol Violation | 5 | 2
Not completed — Other | 6 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Treatment completed, no follow-up | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Extension Phase (Weeks 24 to 52)
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Started | 60 (Number started is different to number completed maintenance phase owing to drop outs (80 subjects).) | 52 (Number started is different to number completed maintenance phase owing to drop outs (85 subjects).)
Completed | 50 | 47
Not Completed | 10 | 5
Not completed — Other | 4 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OROS Hydromorphone HCl | Oxycodone | Total
Number analyzed (Participants) | 254 | 250 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.06) | 58.0 (12.82) | 57.5 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 152 | 294
  Male | 112 | 98 | 210
Region of Enrollment [Number; unit: participants]
  Czech Republic | 34 | 18 | 52
  Denmark | 19 | 20 | 39
  France | 22 | 18 | 40
  Germany | 83 | 80 | 163
  Italy | 17 | 21 | 38
  Norway | 18 | 18 | 36
  Poland | 28 | 34 | 62
  Slovakia | 11 | 11 | 22
  Slovenia | 3 | 5 | 8
  Sweden | 14 | 19 | 33
  Switzerland | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Questionnaire Item 6 "Pain Right Now" Score at Week 24 (Per Protocol [PP] Population)
Description: Assessment of non-inferiority of OROS hydromorphone compared with sustained release (SR) oxycodone with regard to pain control by measuring the change from baseline in pain severity, using BPI item 6 "pain right now" score at week 24. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain right now".
Time Frame: baseline and week 24
Population: PP population (all randomized subjects who took the study medication at least once, who had post-baseline efficacy data, and who were without major protocol violation)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 115 | 108
Units on a scale | -2.8 (2.04) | -3.2 (2.24)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Null hypothesis: Difference in change from baseline with OROS hydromorphone compared with SR oxycodone was less than or equal to 1. Alternative hypothesis: Difference in change from baseline with OROS hydromorphone compared with SR oxycodone was greater than 1. Sample size needed to detect a clinically significant difference of 1 was 151 per treatment arm (standard deviation = 2.4, significance level 0.025 one-sided, based on 90% power); Test type: Non-Inferiority or Equivalence — Tested using 95% confidence interval approach. The non-inferiority margin was 1; p = 0.011, ANCOVA — Statistical significance level was 0.05. Two-sided 95% CI of the treatment difference based on LS means & error terms obtained from ANCOVA (covariate: baseline; factors: country, previous pain treatment, underlying disease, and treatment); If the right side of CI<1 then the null hypothesis was rejected in favour of the alternative, and non-inferiority of OROS hydromorphone was concluded; Mean Difference (Net) = 0.29, 95% CI [-0.27 to 0.84] — LS mean difference has been presented, which was calculated as hydromorphone minus oxycodone

2. Secondary Outcome: Change From Baseline in BPI Pain Severity Sub-score "Pain at Its Worst" (BPI Item 3) at Week 24 (ITT Population)
Description: Change from baseline to week 24 in BPI pain severity, pain at its worst (BPI item 3) assessed using the BPI questionnaire. Score values ranges from 0 (no pain) to 10 (pain as bad as you can imagine). Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain at its worst".
Time Frame: baseline and week 24
Population: ITT population (all randomized subjects who took the study medication at least once, excluding subjects who had no post-baseline efficacy data)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.9 (2.20) | -1.9 (2.24)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Null hypothesis: Difference in change from baseline between hydromorphone and oxycodone was equal to zero. Alternative hypothesis: Difference in change from baseline between hydromorphone and oxycodone was not equal to zero; Test type: Superiority or Other; p = 0.706, ANCOVA — A two-sided significance level of 0.05 was used. A closed hierarchical testing procedure was used to control the overall Type I error. Procedure was stopped here, subsequent tests were exploratory in nature; Superiority of OROS hydromorphone compared to SR oxycodone was evaluated; Mean Difference (Net) = 0.08, 95% CI [-0.32 to 0.47] — Mean difference calculated: hydromorphone minus oxycodone

3. Primary Outcome: Change From Baseline in BPI Questionnaire Item 6 "Pain Right Now" Score at Week 24 (Intent to Treat [ITT] Population)
Description: Assessment of non-inferiority of OROS hydromorphone compared with SR oxycodone with regard to pain control by measuring the change from baseline in pain severity, using BPI item 6 "pain right now" score at week 24. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain right now".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 233 | 223
Units on a scale | -2.1 (2.43) | -2.1 (2.41)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Tested using 95% confidence interval approach. The non-inferiority margin was 1; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.12, 95% CI [-0.53 to 0.29] — Mean difference calculated: hydromorphone minus oxycodone

4. Secondary Outcome: Change From Baseline in Sleep Quality at Week 24
Description: Change from baseline in sleep quality was assessed using the Medical Outcomes Study (MOS) questionnaire at week 24, specifically the sleep subscale index I. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improved sleep quality.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -8.8 (18.44) | -6.2 (18.33)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.065, ANCOVA — A two-sided significance level of 0.05 was used. A closed hierarchical testing procedure was used to control the overall Type I error. Procedure has been stopped, test is exploratory in nature; Superiority of OROS hydromorphone compared to SR oxycodone was evaluated; Mean Difference (Net) = -2.87, 95% CI [-5.94 to 0.19] — Mean difference calculated: hydromorphone minus oxycodone

5. Secondary Outcome: Change From Baseline in Subject Diary Evening Mean Pain Score "Pain Right Now" at Week 24
Description: Change from baseline to week 24 in subject diary evening mean pain score "pain right now". Subjects rated the severity of "pain right now" on a 10 point numeric scale, with 0 being the least pain and 10 being the most pain. Negative change from baseline scores indicate improvement in subject diary evening mean pain score "pain right now".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -2.2 (2.08) | -2.0 (2.33)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.348, ANCOVA — A two-sided significance level of 0.05 was used. A closed hierarchical testing approach was used to control the overall Type I error. Procedure has been stopped, test is exploratory in nature; Superiority of OROS hydromorphone compared to SR oxycodone was evaluated; Mean Difference (Net) = -0.20, 95% CI [-0.62 to 0.22] — Mean difference was calculated: hydromorphone minus oxycodone

6. Secondary Outcome: Change From Baseline in Subject Diary Morning Mean Pain Score "Pain Right Now" at Week 24
Description: Change from baseline to week 24 in subject diary morning mean pain score "pain right now". Subjects rated the severity of "pain right now" on a 10 point numeric scale, with 0 being the least pain and 10 being the most pain. Negative change from baseline scores indicate improvement in subject diary evening mean pain score "pain right now".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -2.0 (2.33) | -2.0 (2.20)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.616, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Superiority of OROS hydromorphone compared to SR oxycodone was evaluated; Mean Difference (Net) = -0.11, 95% CI [-0.54 to 0.32] — Mean difference was calculated: hydromorphone minus oxycodone

7. Secondary Outcome: Number of Subjects With Dose Escalation
Description: Number of subjects with dose increase in study medication.
Time Frame: week 4 and week 24
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 203 | 182
Subjects
  Yes | 27 | 34
  No | 176 | 148
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Null hypothesis: There is no association between study medication and dose escalation. Alternative hypothesis: There is an association between study medication and dose escalation; Test type: Superiority or Other; p = 0.249, Cochran-Mantel-Haenszel — A two-sided significance level of 0.05 was used. A closed hierarchical testing approach was used to control the overall Type I error. Hierarchical testing procedure has been stopped, test is exploratory in nature; Cochran-Mantel-Haenszel Chi-squared statistic stratified for country was used

8. Secondary Outcome: Change From Baseline in BPI Severity Score "Pain Right Now" (BPI Item 6) at Week 4
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "pain right now" (BPI item 6) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain right now".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -2.2 (2.34) | -2.6 (2.26)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.050, ANCOVA — 0.05 two-sided testing, exploratory comparison; Mean Difference (Net) = 0.42, 95% CI [-0.00 to 0.84] — Mean difference calculated: hydromorphone minus oxycodone

9. Secondary Outcome: Change From Baseline in BPI Pain Severity Score "Pain at Its Least" (BPI Item 4) at Week 4
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "pain at its least" (BPI item 4) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain at its least".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.3 (2.03) | -1.8 (2.33)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.105, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.30, 95% CI [-0.06 to 0.67] — Mean difference calculated: hydromorphone minus oxycodone

10. Secondary Outcome: Change From Baseline in BPI Pain Severity "Pain at Its Worst" (BPI Item 3) at Week 4
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "pain at its worst" (BPI item 3) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain at its worst".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.8 (2.14) | -2.1 (1.98)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.058, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.39, 95% CI [-0.01 to 0.79] — Mean difference calculated: hydromorphone minus oxycodone

11. Secondary Outcome: Change From Baseline in BPI Pain Severity "Average Pain" (BPI Item 5) at Week 4
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "average pain" (BPI item 5) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "average pain".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.9 (1.89) | -2.1 (2.10)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.210, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.23, 95% CI [-0.13 to 0.59] — Mean difference calculated: hdromorphone minus oxycodone

12. Secondary Outcome: Change From Baseline in BPI Pain Relief Score (BPI Item 8) at Week 4
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically pain relief (BPI item 8) at week 4. Scores could have ranged from 0 to 100, where 0 = no relief and 100 = complete relief. Positive change from baseline scores indicate improvement in pain relief.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 13.8 (25.15) | 15.2 (26.27)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.941, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.18, 95% CI [-4.87 to 4.52] — Mean difference calculated: hydromorphone minus oxycodone

13. Secondary Outcome: Change From Baseline in BPI Pain Severity Score (Mean of BPI Items 3 to 6) at Week 4
Description: Change from baseline in BPI pain severity was assessed using the BPI questionnaire (mean of BPI items 3 to 6) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in pain severity.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.7 (1.76) | -2.0 (1.90)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.073, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.31, 95% CI [-0.03 to 0.65] — Mean difference calculated: hydromorphone minus oxycodone

14. Secondary Outcome: Change From Baseline in BPI Pain Severity "Pain at Its Least" (BPI Item 4) at Week 24
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "pain at its least" (BPI item 4) at week 24. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain at its least".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.3 (2.23) | -1.4 (2.36)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.431, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.15, 95% CI [-0.52 to 0.22] — Mean difference calculated: hydromorphone minus oxycodone

15. Secondary Outcome: Change From Baseline in BPI Pain Severity "Average Pain" (BPI Item 5) at Week 24
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically "average pain" (BPI item 5) at week 24. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "average pain".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.8 (2.07) | -1.7 (2.22)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.835, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.04, 95% CI [-0.40 to 0.33] — Mean difference calculated: hydromorphone minus oxycodone

16. Secondary Outcome: Change From Baseline in BPI Pain Relief Score (BPI Item 8) at Week 24
Description: Change from baseline in pain severity was assessed using the BPI questionnaire, specifically pain relief (BPI item 8) at week 24. Scores could have ranged from 0 to 100, where 0 = no relief and 100 = complete relief. Positive change from baseline scores indicate improvement in pain relief.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 8.6 (29.32) | 11.5 (28.95)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.837, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.51, 95% CI [-5.36 to 4.35] — Mean difference calculated: hydromorphone minus oxycodone

17. Secondary Outcome: Change From Baseline in BPI Pain Severity Score (Mean of BPI Items 3 to 6) at Week 24
Description: Change in pain severity was assessed using the BPI questionnaire, specifically average (mean) score of BPI items 3 to 6 (worst pain, least pain, average pain, and pain right now) at week 24. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative scores indicate improvement in pain severity.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.6 (1.91) | -1.7 (2.05)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.832, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.04, 95% CI [-0.38 to 0.31] — Mean difference calculated: hydromorphone minus oxycodone

18. Secondary Outcome: Change From Baseline in BPI Interference Score "Interfered With General Activity" (BPI Item 9a) at Week 4
Description: Change from baseline in interference of pain was assessed using the BPI questionnaire, specifically BPI item 9a "pain interfered with general activity" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with general activity".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.6 (2.14) | -1.9 (2.25)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.143, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.30, 95% CI [-0.10 to 0.71] — Mean difference calculated: hydromorphone minus oxycodone

19. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Mood" (BPI Item 9b) at Week 4
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9b "pain interfered with mood" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with mood".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.7 (2.32) | -1.9 (2.57)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.345, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.21, 95% CI [-0.23 to 0.64] — Mean difference calculated: hydromorphone minus oxycodone

20. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Walking Ability" (BPI Item 9c) at Week 4
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9c "pain interfered with walking ability" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with walking ability".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.2 (2.63) | -1.5 (2.63)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.552, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.14, 95% CI [-0.33 to 0.61] — Mean difference calculated: hydromorphone minus oxycodone

21. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Normal Work" (BPI Item 9d) at Week 4
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9d "pain interfered with normal work" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with normal work".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.4 (2.40) | -2.0 (2.70)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.042, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.47, 95% CI [0.02 to 0.93] — Mean difference calculated: hydromorphone minus oxycodone

22. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Relations With Other People" (BPI Item 9e) at Week 4
Description: Change from baseline in pain interference was assessed using BPI questionnaire, specifically BPI item 9e "pain interfered with relations with other people" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with relations with other people".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.1 (2.56) | -1.4 (2.95)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.171, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.33, 95% CI [-0.14 to 0.81] — Mean difference calculated: hydromorphone minus oxycodone

23. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Sleep" (BPI Item 9f) at Week 4
Description: Change from baseline in pain interference was assessed using BPI questionnaire, specifically BPI item 9f "pain interfered with sleep" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 - completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with sleep".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -2.1 (2.34) | -2.3 (3.07)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.475, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.17, 95% CI [-0.31 to 0.65] — Mean difference calculated: hydromorphone minus oxycodone

24. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Enjoyment of Life" (BPI Item 9g) at Week 4
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9g "pain interfered with enjoyment of life" at week 4. Scores could have ranged from 0 to 10, where 0 = does not interfere and 10 = interferes completely. Negative change from baseline scores indicate improvement in "pain interfered with enjoyment of life".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.6 (2.62) | -1.9 (2.97)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.359, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.23, 95% CI [-0.26 to 0.72] — Mean difference calculated: hydromorphone minus oxycodone

25. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With General Activity" (BPI Item 9a) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9a "pain interfered with general activity" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with general activity".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.6 (2.42) | -1.6 (2.46)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.611, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.11, 95% CI [-0.52 to 0.30] — Mean difference calculated: hydromorphone minus oxycodone

26. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Mood" (BPI Item 9b) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9b "pain interfered with mood" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with mood".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.4 (2.85) | -1.3 (2.88)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.526, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.15, 95% CI [-0.60 to 0.31] — Mean difference calculated: hydromorphone minus oxycodone

27. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Walking Ability" (BPI Item 9c) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9c "pain interfered with walking ability" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with walking ability".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.1 (2.75) | -1.2 (2.51)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.769, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.06, 95% CI [-0.49 to 0.36] — Mean difference calculated: hydromorphone minus oxycodone

28. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Normal Work" (BPI Item 9d) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9d "pain interfered with normal work" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with normal work".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.3 (2.63) | -1.4 (2.68)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.843, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.04, 95% CI [-0.40 to 0.49] — Mean difference calculated: hydromorphone minus oxycodone

29. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Relations With Other People" (BPI Item 9e) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9e "pain interfered with relations with other people" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with relations with other people".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -0.7 (2.92) | -0.9 (2.75)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.977, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.01, 95% CI [-0.45 to 0.44] — Mean difference calculated: hydromorphone minus oxycodone

30. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Sleep" (BPI Item 9f) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9f "pain interfered with sleep" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with sleep".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.4 (2.76) | -1.5 (3.08)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.977, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 0.01, 95% CI [-0.47 to 0.49] — Mean difference calculated: hydromorphone minus oxycodone

31. Secondary Outcome: Change From Baseline in Pain Interference "Pain Interfered With Enjoyment of Life" (BPI Item 9g) at Week 24
Description: Change from baseline in pain interference was assessed using the BPI questionnaire, specifically BPI item 9g "pain interfered with enjoyment of life" at week 24. Scores could have ranged from 0 to 10, where 0 = does not interfere to 10 = completely interferes. Negative change from baseline scores indicate improvement in "pain interfered with enjoyment of life".
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.2 (2.91) | -1.3 (3.09)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.902, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.03, 95% CI [-0.51 to 0.45] — Mean difference calculated: hydromorphone minus oxycodone

32. Secondary Outcome: Change From Baseline in BPI Pain Severity, Relief and Interference Scores (Extension Phase)
Description: Change from baseline in pain severity, pain relief, and pain interference was assessed using the BPI questionnaire at week 52. BPI items 3 to 6, score range 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine; BPI items 9a to 9g, score range from 0 to 10, where 0 = does not interfere and 10 = completely interferes. Negative change from baseline scores indicate improvement in pain severity and pain interference. BPI item 8, score range from 0 to 100, where 0 = no relief and 100 = complete relief. Positive change from baseline scores indicate improvement in pain relief.
Time Frame: baseline and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale
  Pain severity, BPI items 3 to 6 | -2.4 (1.67) | -2.4 (2.13)
  Pain relief, BPI item 8 | 17.7 (26.36) | 23.6 (25.46)
  Pain right now, BPI item 6 | -2.9 (2.07) | -2.8 (2.16)
  Pain at its worst, BPI item 3 | -2.8 (2.07) | -2.4 (2.29)
  Pain at its least, BPI item 4 | -1.9 (2.14) | -2.3 (2.59)
  Average pain, BPI item 5 | -2.6 (1.78) | -2.6 (2.21)
  Pain interfered general activity, BPI item 9a | -2.5 (2.28) | -2.6 (2.40)
  Pain interfered mood, BPI item 9b | -2.3 (2.42) | -2.7 (3.12)
  Pain interfered walking ability, BPI item 9c | -2.3 (2.10) | -2.5 (2.89)
  Pain interfered normal work, BPI item 9d | -2.9 (2.64) | -3.2 (2.63)
  Pain interfered relation other people, BPI item 9e | -1.6 (2.56) | -1.9 (3.34)
  BPI pain interfered sleep, BPI item 9f | -2.4 (2.61) | -3.0 (3.02)
  BPI pain interfered enjoyment of life, BPI item 9g | -2.4 (2.63) | -2.6 (3.32)

33. Secondary Outcome: Change From Baseline in Sleep Quality (MOS Index I) at Week 4
Description: Change from baseline in sleep quality was assessed using the sleep subscales of the MOS questionnaire, which consists of 12 items; MOS sleep scale index I (average of item 1, 3, 7, 8, 9, and 12) was assessed at week 4. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep quality.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -10.6 (17.61) | -8.7 (18.83)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.169, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -2.36, 95% CI [-5.74 to 1.02] — Mean difference calculated: hydromorphone minus oxycodone

34. Secondary Outcome: Change From Baseline in Sleep Quality (MOS Index II) at Week 4
Description: Change from baseline in sleep quality was assessed using the sleep subscales of the MOS questionnaire, which consists of 12 items. MOS index II (average of items 1, 3, 4, 5, 6, 7, 8, 9, and 12) was assessed at week 4. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep quality.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -10.5 (16.40) | -9.0 (17.80)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.245, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -1.89, 95% CI [-5.09 to 1.31] — Mean difference calculated: hydromorphone minus oxycodone

35. Secondary Outcome: Change From Baseline in Sleep Quality (MOS Index II) at Week 24
Description: Change from baseline in sleep quality was assessed using the sleep subscales of the MOS questionnaire, which consists of 12 items. MOS index II (average of items 1, 3, 4, 5, 6, 7, 8, 9, and 12) was assessed at week 24. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep quality.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -8.9 (17.28) | -6.5 (16.73)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.071, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -2.64, 95% CI [-5.51 to 0.23] — Mean difference calculated: hydromorphone minus oxycodone

36. Secondary Outcome: Change From Baseline in Sleep Quality, Sleep Disturbance at Week 24
Description: Change from baseline in sleep quality (sleep disturbance) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep disturbance.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -13.1 (22.77) | -11.7 (22.95)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.297, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -2.03, 95% CI [-5.85 to 1.80] — Mean difference calculated: hydromorphone minus oxycodone

37. Secondary Outcome: Change From Baseline in Sleep Quality, Snoring at Week 24
Description: Change from baseline in sleep quality (snoring) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in snoring.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.0 (22.04) | -4.1 (21.93)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.205, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 2.41, 95% CI [-1.32 to 6.14] — Mean difference calculated: hydromorphone minus oxycodone

38. Secondary Outcome: Change From Baseline in Sleep Quality, Sleep Shortness of Breath or Headache at Week 24
Description: Change from baseline in sleep quality (sleep shortness of breath or headache) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep shortness of breath or headache.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -5.3 (28.44) | -0.1 (24.27)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.107, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -3.35, 95% CI [-7.43 to 0.73] — Mean difference calculated: hydromorphone minus oxycodone

39. Secondary Outcome: Change From Baseline in Sleep Quality, Sleep Adequacy at Week 24
Description: Change from baseline in sleep quality (sleep adequacy) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = worst sleep quality and 100 = best sleep quality. Positive change from baseline scores indicate improvement in sleep adequacy.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 9.1 (28.10) | 7.3 (26.63)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.475, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = 1.60, 95% CI [-2.80 to 6.00] — Mean difference calculated: hydromorphone minus oxycodone

40. Secondary Outcome: Change From Baseline in Sleep Quality, Sleep Somnolence at Week 24
Description: Change from baseline in sleep quality (sleep somnolence) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = best sleep quality and 100 = worst sleep quality. Negative change from baseline scores indicate improvement in sleep somnolence.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -1.6 (21.70) | 3.0 (20.91)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.020, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -4.16, 95% CI [-7.67 to -0.65] — Mean difference calculated: hydromorphone minus oxycodone

41. Secondary Outcome: Change From Baseline in Sleep Quality, Sleep Quantity at Week 24
Description: Change from baseline in sleep quality (sleep quantity) was assessed using the MOS questionnaire at week 24. Score range 0 to 100, where 0 = worst sleep quality and 100 = best sleep quality. Positive change from baseline scores indicate improvement in sleep quantity.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 0.4 (1.86) | 0.5 (1.51)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.880, ANCOVA — 0.05 two-sided test; Mean Difference (Net) = -0.02, 95% CI [-0.30 to 0.26] — Mean difference calculated: hydromorphone minus oxycodone

42. Secondary Outcome: Number of Subjects Indicating That They Had Optimal Sleep at Week 24
Description: Number of subjects indicating that they had optimal sleep was assessed based on the number of hours of sleep reported on the MOS questionnaire at week 24. Optimal sleep was defined as 7 to 8 hours sleep per night.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 249 | 242
Subjects
  Yes | 83 | 71
  No | 166 | 171
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.320, Cochran-Mantel-Haenszel

43. Secondary Outcome: Change From Baseline in Sleep Quality at Week 52
Description: Change from baseline in sleep quality was assessed using the MOS questionnaire at week 52. Score range 0 to 100. For disturbance, snoring, shortness of breath or headache, and somnolence, 0 = best sleep quality and 100 = worst sleep quality; negative change from baseline scores indicate improvement in sleep quality for these measures. For adequacy and quantity, 0 = worst sleep quality and 100 = best sleep quality; positive change from baseline scores indicate improvement in sleep quality for these measures.
Time Frame: baseline and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale
  MOS sleep disturbance | -17.6 (22.44) | -20.1 (23.17)
  MOS snoring | -2.5 (23.01) | -4.7 (23.86)
  MOS sleep shortness of breath or headache | -8.4 (19.89) | -7.8 (21.94)
  MOS sleep adequacy | 12.3 (27.06) | 11.9 (30.74)
  MOS sleep somnolence | -6.5 (20.49) | 1.8 (21.54)
  MOS sleep quantity | 0.5 (2.27) | 0.5 (1.25)

44. Secondary Outcome: Number of Subjects Indicating Optimal Sleep at Week 52
Description: Number of subjects who experienced optimal sleep was assessed based on the number of hours of sleep reported on the MOS questionnaire at week 52. Optimal sleep was defined as 7-8 hours sleep per night.
Time Frame: week 52
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 55 | 49
Subjects
  Yes | 27 | 19
  No | 28 | 30

45. Secondary Outcome: Change From Baseline in Subject Diary Mean Pain Evening, Morning, and All Day Scores at Week 24
Description: Change from baseline to week 24 in subject diary evening, morning and all day mean pain scores for pain right now, at its worst, at its least, and average. Subjects rated the severity of pain on a 10 point numeric scale, with 0 being the least pain and 10 being the most pain. Negative change from baseline scores indicate improvement in subject diary mean pain scores.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale
  Evening worst pain | -2.2 (2.32) | -2.1 (2.31)
  Evening least pain | -1.6 (2.28) | -1.4 (2.36)
  Evening average pain | -2.0 (2.12) | -1.8 (2.22)
  Morning worst pain | -1.9 (2.38) | -2.1 (2.34)
  Morning least pain | -1.5 (2.44) | -1.2 (2.44)
  Morning average pain | -1.7 (2.20) | -1.8 (2.30)
  All day worst pain | -2.1 (2.11) | -2.1 (2.09)
  All day least pain | -1.5 (2.21) | -1.3 (2.22)
  All day average pain | -1.8 (2.00) | -1.8 (2.08)
  All day pain right now | -2.1 (2.05) | -2.0 (2.20)

46. Secondary Outcome: Change From Baseline in Subject Diary Mean Pain Score for "Pain at Its Worst" From Morning to Evening at Weeks 4, 8, 12, 16, 20, and 24
Description: Change from baseline in subject diary mean pain score "pain at its worst" from morning to evening at weeks 4, 8, 12, 16, 20, and 24. Subjects rated the severity of "pain right now" on a 10 point numeric scale, with 0 being the least pain and 10 being the most pain. Negative change from baseline scores indicate improvement in subject diary mean pain score "pain at its worst".
Time Frame: baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale
  Baseline | 0.7 (1.93) | 0.4 (1.88)
  Week 4 | 0.5 (1.30) | 0.4 (1.22)
  Week 8 | 0.4 (1.23) | 0.4 (1.42)
  Week 12 | 0.3 (1.23) | 0.3 (1.26)
  Week 16 | 0.2 (1.08) | 0.2 (1.28)
  Week 20 | 0.3 (1.13) | 0.2 (1.14)
  Week 24 | 0.3 (1.23) | 0.3 (1.07)

47. Secondary Outcome: Number of Subjects With Dose Escalation at Week 4 (ITT Population)
Description: The number of subjects with dose increase in study medication was assessed at week 4.
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  Yes | 175 | 166
  No | 79 | 84
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.575, Cochran-Mantel-Haenszel

48. Secondary Outcome: Number of Subjects With Dose Escalation at Week 24 (ITT Population)
Description: The number of subjects with dose increase in study medication was assessed at week 24.
Time Frame: week 24
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 203 | 182
Subjects
  Yes | 146 | 145
  No | 57 | 37
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.807, Cochran-Mantel-Haenszel

49. Secondary Outcome: Change From Baseline in Quality of Life (QoL) "Bodily Pain" at Week 4
Description: Change from baseline in QoL was assessed using the Short Form (SF)-36 QoL questionnaire, specifically the SF-36 bodily pain index. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in bodily pain.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 13.7 (18.10) | 16.7 (18.43)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.118, ANCOVA; Mean Difference (Net) = -2.61, 95% CI [-5.88 to 0.67] — Mean difference calculated: hydromorphone minus oxycodone

50. Secondary Outcome: Change From Baseline in QoL "General Health Perceptions" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 general health perceptions score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in general health perceptions.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 3.9 (14.43) | 5.0 (16.97)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.956, ANCOVA; Mean Difference (Net) = -0.08, 95% CI [-3.08 to 2.91] — Mean difference calculated: hydromorphone minus oxycodone

51. Secondary Outcome: Change From Baseline in QoL "Health Transition" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 health transition score at week 4. Scores could range from 0 to 100, with higher scores indicating a better QoL. Positive change from baseline scores indicate improvement in health transition.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -0.4 (1.08) | -0.5 (0.99)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.299, ANCOVA; Mean Difference (Net) = 0.09, 95% CI [-0.08 to 0.26] — Mean difference calculated: hydromorphone minus oxycodone

52. Secondary Outcome: Change From Baseline in QoL "Mental Health" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 mental health score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in mental health score.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 6.2 (15.76) | 6.6 (17.17)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.471, ANCOVA; Mean Difference (Net) = -1.13, 95% CI [-4.20 to 1.95] — Mean difference calculated: hydromorphone minus oxymorphone

53. Secondary Outcome: Change From Baseline in QoL "Physical Functioning" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 physical functioning score at week 4. Scores could range from 0 to 100, with high scores indicating a better QoL. Positive change from baseline scores indicate improvement in physical functioning.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 8.7 (17.05) | 5.4 (16.80)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.025, ANCOVA; Mean Difference (Net) = 3.84, 95% CI [0.48 to 7.19] — Mean difference calculated: hydromorphone minus oxycodone

54. Secondary Outcome: Change From Baseline in QoL "Role Emotional" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 "role emotional" score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in "role emotional".
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 9.9 (43.25) | 4.7 (48.03)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.556, ANCOVA; Mean Difference (Net) = 2.40, 95% CI [-5.61 to 10.42] — Mean difference calculated: hydromorphone minus oxycodone

55. Secondary Outcome: Change From Baseline in QoL "Role Physical" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 role physical score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in role physical.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 13.2 (36.84) | 16.9 (36.08)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.551, ANCOVA; Mean Difference (Net) = -2.12, 95% CI [-9.11 to 4.88] — Mean difference calculated: hydromorphone minus oxycodone

56. Secondary Outcome: Change From Baseline in QoL "Social Functioning" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 social functioning score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in social functioning.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 10.5 (25.33) | 12.9 (26.39)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.207, ANCOVA; Mean Difference (Net) = -2.98, 95% CI [-7.63 to 1.66] — Mean difference calculated: hydromorphone minus oxycodone

57. Secondary Outcome: Change From Baseline in QoL "Vitality" at Week 4
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 vitality score at week 4. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in vitality.
Time Frame: baseline and week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 6.4 (16.92) | 9.2 (17.08)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.123, ANCOVA; Mean Difference (Net) = -2.46, 95% CI [-5.60 to 0.68] — Mean difference calculated: hydromorphone minus oxycodone

58. Secondary Outcome: Change From Baseline in QoL "Bodily Pain" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 bodily pain index score at week 24. Score could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in bodily pain.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 10.6 (21.04) | 11.9 (19.83)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.602, ANCOVA; Mean Difference (Net) = -0.90, 95% CI [-4.27 to 2.48] — Mean difference calculated: hydromorphone minus oxycodone

59. Secondary Outcome: Change From Baseline in QoL "General Health Perceptions" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 general health perceptions at week 24. Scores could range from 0 to 100 with a higher score indicating a better QoL. Positive change from baseline scores indicate improvement in health perceptions.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 2.1 (17.04) | 2.2 (16.61)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.647, ANCOVA; Mean Difference (Net) = 0.65, 95% CI [-2.14 to 3.44] — Mean difference calculated: hydromorphone minus oxycodone

60. Secondary Outcome: Change From Baseline in QoL "Health Transition" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 health transition score at week 24. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in health transition.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | -0.2 (1.03) | -0.1 (0.96)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.627, ANCOVA; Mean Difference (Net) = -0.03, 95% CI [-0.17 to 0.10] — Mean difference calculated: hydromorphone minus oxycodone

61. Secondary Outcome: Change From Baseline in QoL "Mental Health" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 mental health score at week 24. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline score indicates improvement in mental health.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 2.6 (19.30) | 2.6 (18.79)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.414, ANCOVA; Mean Difference (Net) = -1.30, 95% CI [-4.45 to 1.84] — Mean difference calculated: hydromorphone minus oxycodone

62. Secondary Outcome: Change From Baseline in QoL "Physical Functioning" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 physical functioning score at week 24. Scores could range from 0 to 100, with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in physical functioning.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 7.7 (19.09) | 4.4 (15.33)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Net) = 4.05, 95% CI [0.94 to 7.16] — Mean difference calculated: hydromorphone minus oxycodone

63. Secondary Outcome: Change From Baseline in QoL "Role Emotional" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 "role emotional" score at week 24. Scores could range from 0 to 100 with a higher score indicating a better QoL. Positive change from baseline scores indicate improvement in "role emotional."
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 0.40 (47.71) | -1.5 (47.22)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.955, ANCOVA; Mean Difference (Net) = 0.21, 95% CI [-7.20 to 7.62] — Mean difference calculated: hydromorphone minus oxycodone

64. Secondary Outcome: Change From Baseline in QoL "Role Physical" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 role physical score at week 24. Scores could range from 0 to 100 with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in role physical.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 8.8 (37.80) | 9.9 (34.11)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.669, ANCOVA; Mean Difference (Net) = 1.31, 95% CI [-4.72 to 7.34] — Mean difference calculated: hydromorphone minus oxycodone

65. Secondary Outcome: Change From Baseline in QoL "Social Functioning" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 social functioning score at week 24. Scores could range from 0 to 100 with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in social functioning.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 6.6 (27.81) | 5.0 (26.85)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.595, ANCOVA; Mean Difference (Net) = 1.17, 95% CI [-3.15 to 5.49] — Mean difference calculated: hydromorphone minus oxycodone

66. Secondary Outcome: Change From Baseline in QoL "Vitality" at Week 24
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire, specifically SF-36 vitality score at week 24. Scores could range from 0 to 100 with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in vitality.
Time Frame: baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale | 4.3 (19.73) | 5.6 (17.93)
Statistical Analysis 1: Comparison: OROS Hydromorphone HCl vs Oxycodone; Exploratory comparison; Test type: Superiority or Other; p = 0.543, ANCOVA; Mean Difference (Net) = -0.94, 95% CI [-3.98 to 2.10] — Mean difference calculated: hydromorphone minus oxycodone

67. Secondary Outcome: Change From Baseline in QoL at Week 52
Description: Change from baseline in QoL was assessed using the SF-36 QoL questionnaire at week 52. Scores could range from 0 to 100 with a high score indicating a better QoL. Positive change from baseline scores indicate improvement in QoL.
Time Frame: baseline and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Units on a scale
  SF-36 bodily pain index | 23.1 (22.07) | 19.6 (22.67)
  SF-36 general health perceptions | 9.6 (17.86) | 5.5 (18.97)
  SF-36 health transition | -0.3 (0.90) | -0.1 (1.03)
  SF-36 mental health | 11.7 (17.21) | 6.9 (26.03)
  SF-36 physical functioning | 11.4 (20.10) | 9.2 (20.12)
  SF-36 role emotional | 22.1 (48.86) | 7.3 (56.86)
  SF-36 role physical | 17.0 (38.02) | 15.0 (33.50)
  SF-36 social functioning | 15.4 (23.11) | 12.8 (28.29)
  SF-36 vitality | 11.5 (17.39) | 11.9 (21.40)

68. Secondary Outcome: Clinical Global Assessment of Efficacy
Description: Overall clinical efficacy was assessed by the Investigator using the following global ratings: very good, good, moderate, poor, or very poor, at weeks 4, 24, and 52.
Time Frame: weeks 4, 24, and 52
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  Visit 5, week 4: very good | 49 | 27
  Visit 5, week 4: good | 92 | 92
  Visit 5, week 4: moderate | 51 | 50
  Visit 5, week 4: poor | 12 | 9
  Visit 5, week 4: very poor | 0 | 3
  Visit 8, week 24: very good | 48 | 31
  Visit 8, week 24: good | 91 | 103
  Visit 8, week 24: moderate | 50 | 41
  Visit 8, week 24: poor | 44 | 50
  Visit 8, week 24: very poor | 16 | 10
  Visit 10, week 52: very good | 18 | 11
  Visit 10, week 52: good | 37 | 34
  Visit 10, week 52: moderate | 5 | 6
  Visit 10, week 52: poor | 0 | 1
  Visit 10, week 52: very poor | 0 | 0

69. Secondary Outcome: Change in Dose of Study Treatment
Description: Number of subjects with change in dose of study treatment was assessed at weeks 4, 24, and 52.
Time Frame: weeks 4, 24, and 52
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  0 mg (week 4) | 79 | 84
  +8 mg (week 4) | 102 | 0
  +20 mg (week 4) | 0 | 108
  +24 mg (week 4) | 73 | 0
  +60 mg (week 4) | 0 | 58
  -60 mg (week 24) | 0 | 2
  -40 mg (week 24) | 0 | 8
  -24 mg (week 24) | 1 | 0
  -20 mg (week 24) | 0 | 6
  -16 mg (week 24) | 4 | 0
  -8 mg (week 24) | 11 | 0
  0 mg (week 24) | 172 | 144
  +8 mg (week 24) | 6 | 0
  +16 mg (week 24) | 9 | 0
  +20 mg (week 24) | 0 | 8
  +40 mg (week 24) | 0 | 14
  -16 mg (week 52) | 3 | 0
  -8 mg (week 52) | 1 | 0
  0 mg (week 52) | 56 | 50
  +40 mg (week 52) | 0 | 2

70. Secondary Outcome: Change in Dose of Study Treatment During Titration Phase (First 4 Weeks of Study) and Overall Treatment Phase I (First 24 Weeks of Study)
Description: Number of subejcts with change in dose of study treatment was assessed and stratified by time on study, at least 4 weeks versus dropped out at highest dose before week 4, at weeks 4 and 24.
Time Frame: weeks 4 and 24
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  Titration phase (on study at least 4 weeks) 0 mg | 50 | 41
  Titration phase (on study at least 4 weeks) +8 mg | 92 | 0
  Titration phase (on study at least 4 weeks) +20 mg | 0 | 94
  Titration phase (on study at least 4 weeks) +24 mg | 65 | 0
  Titration phase (on study at least 4 weeks) +60 mg | 0 | 54
  Titration phase (on study <4 weeks) 0 mg | 29 | 43
  Titration phase (on study <4 weeks) +8 mg | 10 | 0
  Titration phase (on study <4 weeks) +20 mg | 0 | 14
  Titration phase (on study <4 weeks) +24 mg | 8 | 0
  Titration phase (on study <4 weeks) +60 mg | 0 | 4
  Week 24 (on study at least 4 weeks) 0 mg | 58 | 40
  Week 24 (on study at least 4 weeks ) +4 mg | 0 | 1
  Week 24 (on study at least 4 weeks ) +8 mg | 76 | 0
  Week 24 (on study at least 4 weeks) +20 mg | 0 | 87
  Week 24 (on study at least 4 weeks ) +24 mg | 73 | 0
  Week 24 (on study at least 4 weeks) +60 mg | 0 | 61
  Week 24 (on study <4 weeks) 0 mg | 29 | 43
  Week 24 (on study <4 weeks) +8 mg | 10 | 0
  Week 24 (on study <4 weeks) +20 mg | 0 | 14
  Week 24 (on study <4 weeks) +24 mg | 8 | 0
  Week 24 (on study <4 weeks) +60 mg | 0 | 4

71. Secondary Outcome: Number of Drop-outs
Description: Number of drop-outs according to reasons for drop-out and due to inefficacy at maximal dosage was assessed at weeks 24 and 52.
Time Frame: baseline to week 24 (core); week 24 to week 52 (extension)
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  Adverse events (core) | 57 | 56
  Adverse events (extension) | 4 | 1
  Consent withdrawn (core) | 12 | 16
  Consent withdrawn (extension) | 0 | 1
  Inadequate pain relief (core) | 22 | 18
  Inadequate pain relief (extension) | 0 | 1
  Investigator withdrew patient (core) | 4 | 2
  Investigator withdrew patient (extension) | 0 | 0
  Lost to follow up (core) | 2 | 0
  Lost to follow up (extension) | 1 | 0
  Non compliance (core) | 3 | 10
  Non compliance (extension) | 1 | 0
  Other (core) | 6 | 5
  Other (extension) | 4 | 2
  Protocol violation (core) | 6 | 6
  Protocol violation (extension) | 0 | 0
  Treatment completed no follow up visit (core) | 2 | 0
  Treatment completed no follow up visit (extension) | 0 | 0
  Inefficacy at maximal dosage (core) | 17 | 12

72. Secondary Outcome: Number of Days With add-on Pain Medication
Description: Number of days with add-on pain medication during the first 24 weeks of the study was assessed at week 24.
Time Frame: week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Days | 68.2 (59.6) | 66.1 (61.2)

73. Secondary Outcome: Amount of add-on Pain Medication
Description: Total amount of add-on pain medication (paracetamol) for the first 24 weeks was assessed at week 24.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
mg | 80004.8 (97004.53) | 76191.9 (96925.72)

74. Secondary Outcome: Mode and Convenience of Drug Intake.
Description: Subjects filled out a questionnaire based on the mode and convenience of drug intake and could rate their responses as very convenient, convenient, neither convenient or inconvenient, inconvenient, and very inconvenient.
Time Frame: weeks 4, 24, and 52
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Subjects
  Very convenient, week 4 | 57 (0.86) | 36 (0.77)
  Convenient, week 4 | 97 (0.96) | 94 (1.01)
  Neither convenient or inconvenient, week 4 | 30 (0.61) | 30 (0.61)
  Inconvenient, week 4 | 7 | 6
  Very inconvenient, week 4 | 3 | 1
  Very convenient, week 24 | 63 | 53
  Convenient, week 24 | 96 | 90
  Neither convenient or inconvenient, week 24 | 31 | 33
  Inconvenient, week 24 | 8 | 11
  Very inconvenient, week 24 | 7 | 8
  Very convenient, week 52 | 21 | 11
  Convenient, week 52 | 10 | 15
  Neither convenient or inconvenient, week 52 | 2 | 2
  Inconvenient, week 52 | 0 | 0
  Very inconvenient, week 52 | 0 | 0

75. Secondary Outcome: Resource Utilization of Pain Management
Description: Resource utilization was defined as the number of additional visits including additional telephone visits during the treatment period. This was assessed at week 24.
Time Frame: week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Additional visits
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
Additional visits | 2.1 (2.21) | 1.9 (2.29)

76. Primary Outcome: Equi-analgesic Dosage of OROS Hydromorphone Once-daily and SR Oxycodone Twice-daily (PP Population)
Description: If non-inferiority of OROS hydromorphone was established, the daily dose of OROS hydromorphone and SR oxycodone that induced the same pain control was to be calculated (average dose used at week 24). Relative equi-analgesic dose was defined as mean dose/allowed maximum dose*100. Allowed maximum doses were 32mg OROS hydromorphone and 80mg SR oxycodone respectively.
Time Frame: week 24
Population: PP population (all subjects who took the study medication at least once, who had post-baseline efficacy data, and who were without major protocol violation)
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 115 | 108
mg per day | 18.9 (9.44) | 48.3 (22.4)

77. Primary Outcome: Equi-analgesic Dosage of OROS Hydromorphone Once-daily and SR Oxycodone Twice-daily (ITT Population)
Description: as for outcome 76
Time Frame: week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
mg per day | 18.4 (9.92) | 43.8 (23.12)

78. Primary Outcome: Equi-analgesic Dose at Steady-state (PP Population)
Description: Dose of OROS hydromorphone and SR oxycodone that induced the same pain control at steady state, defined as the mean dose from week 4 to week 24.
Time Frame: week 4 to week 24
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 115 | 108
mg per day | 18.95 (9.223) | 47.82 (21.663)

79. Primary Outcome: Equi-analgesic Dose at Steady State (ITT Population)
Description: as for outcome 78
Time Frame: week 4 to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Number analyzed (Participants) | 254 | 250
mg per day | 19.50 (9.584) | 48.41 (21.835)

ADVERSE EVENTS:
Arm/Group | OROS Hydromorphone HCl | Oxycodone
Serious Adverse Events (participants affected / at risk) | 25/254 | 21/250
Other Adverse Events (participants affected / at risk) | 206/254 | 212/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OROS Hydromorphone HCl (N=254) | Oxycodone (N=250)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectocele (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy liver (Investigations) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Pain management (Surgical and medical procedures) | 0 (0) | 1 (1)
Prosthesis implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OROS Hydromorphone HCl (N=254) | Oxycodone (N=250)
Vertigo (Ear and labyrinth disorders) | 14 (14) | 16 (17)
Constipation (Gastrointestinal disorders) | 73 (92) | 65 (76)
Diarrhoea (Gastrointestinal disorders) | 33 (45) | 14 (15)
Nausea (Gastrointestinal disorders) | 68 (82) | 78 (92)
Vomiting (Gastrointestinal disorders) | 32 (38) | 36 (43)
Fatigue (General disorders) | 35 (37) | 31 (33)
Anorexia (Metabolism and nutrition disorders) | 14 (16) | 13 (13)
Dizziness (Nervous system disorders) | 17 (18) | 26 (30)
Headache (Nervous system disorders) | 22 (26) | 25 (32)
Somnolence (Nervous system disorders) | 9 (10) | 18 (23)
Insomnia (Psychiatric disorders) | 13 (13) | 15 (17)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 29 (35) | 22 (22)
Pruritis (Skin and subcutaneous tissue disorders) | 25 (27) | 26 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days